CLINICAL TRIAL: NCT01265147
Title: Phase II Study to Evaluate Efficacy and Safety of Intensity-modulated Radiation Therapy Combined With Cisplatin or Nedaplatin Chemotherapy in Patients With Nasopharyngeal Carcinoma
Brief Title: Intensity-modulated Radiation Therapy Combined With Cisplatin or Nedaplatin Chemotherapy in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Zhenzhou Yang, Daping Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Daping H 001
Record Dates: First submitted 2010-12-03; First posted 2010-12-23 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2010-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cisplatin (Active Comparator): cisplatin combine with IMRT
  Interventions: Drug: Cisplatin
- Nedaplatin (Experimental): Nedaplatin combine with IMRT
  Interventions: Drug: Nedaplatin

INTERVENTIONS:
Drug: Cisplatin — 40mg/m2/w
  Arms: Cisplatin
Drug: Nedaplatin — 40mg/m2/w
  Arms: Nedaplatin

SUMMARY:
This phase II trial is studying cisplatin or nedaplatin combine with IMRT to evaluate which one is better efficacy and security in nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Age≥18,T1-2aN1-3;T2-4NxNPC,VEGFR+,++,KPS>70,Life expectancy≥6 months, No uncontrolled hypertension,cardiac failure,diabetes,lunacy

Exclusion Criteria:

Distant metastasis, recurrent disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
locoregionally control rate | 3 months
  3 months after treatment

SECONDARY OUTCOMES:
Survival | 1,3,5 years
  1 year Progress Free Survival,Disease Free Survival,3 years and 5 years Over All Survival,Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, China